CLINICAL TRIAL: NCT00095446
Title: An Open-Label, Multi Center, Clinical Trial: External Continuous Subcutaneous Infusion of Insulin Using Insulin Aspart (NovoLog®) in Subjects With Type 1 and Insulin Requiring Type 2 Diabetes
Brief Title: NovoLog Observation Trial in Subjects With Type 1 and Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ANA-2190
Record Dates: First submitted 2004-11-04; First posted 2004-11-05 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus; Diabetes
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: insulin aspart

SUMMARY:
This trial is conducted in the United States of America (USA). The aim of this trial is to assess control of blood sugar, safety, and patient acceptance of insulin aspart compared to insulin lispro, both in insulin pumps, in standard clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* People with Type I or Type II Diabetes
* 18 Years or Older.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 513 (Actual)
Dates: Start 2004-07; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Treatment satisfaction with insulin pump therapy

SECONDARY OUTCOMES:
body weight
Insulin dose
Overall glycemic control
number and types of infusion sets used.
infusion set in-use times

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR,1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Princeton, New Jersey, United States

REFERENCES:
- [Result] Wittlin SD, Marcus AO, Weng CS, Howard CP, Schorr AB; CONTROL Study Group. Evaluation of treatment satisfaction associated with the use of insulin aspart in continuous subcutaneous insulin infusion. Diabetes Technol Ther. 2008 Feb;10(1):1-10. doi: 10.1089/dia.2007.0234. PMID 18275357
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com